CLINICAL TRIAL: NCT00813293
Title: Randomized, Double-Blind, Placebo-Controlled, Phase II Trial Of Short Course Sorafenib Therapy Prior to Radiofrequency Ablation for Intermediate Sized (3.5 to 7cm) Hepatocellular Cancer
Brief Title: Sorafenib Therapy Prior to Radiofrequency Ablation for Intermediate Sized Hepatocellular Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Bayer (Industry); Onyx Therapeutics, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Bullock, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-256; K23CA139005 (NIH); IST000508 (Other Grant/Funding Number: Bayer/Onyx)
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatocellular Cancer; HCC; Liver Cancer; radiofrequency ablation; RFA; sorafenib; nexavaar; liver directed therapy; interventional radiology
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Experimental): Participants received a nine-day course of oral sorafenib 400 mg twice a day and radiofrequency ablation (RFA) on Day 10. Tumors in each group underwent RFA using a standard regimen (1 cm tip, 70 ± 2º C, 5 min).
  Interventions: Drug: Sorafenib; Procedure: radiofrequency ablation
- Placebo (Placebo Comparator): Participants received a nine-day course of placebo pills twice a day and radiofrequency ablation (RFA) on Day 10. Tumors in each group underwent RFA using a standard regimen (1 cm tip, 70 ± 2º C, 5 min).
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Drug: Sorafenib
  Other Names: Nexavar
  Arms: Sorafenib
Procedure: radiofrequency ablation
  Other Names: RFA

SUMMARY:
The purpose of this research study is to determine if sorafenib improves the effectiveness of a procedure called radiofrequency ablation (RFA) for the treatment of hepatocellular cancer (HCC). Radiofrequency ablation has been used to treat many types of tumors, including hepatocellular cancers. During RFA a needle is inserted into the tumor tissue and heat is used to kill the tumor cells. Sorafenib has been approved by the FDA for the treatment of hepatocellular cancer that cannot be treated with surgery. Pre-clinical data suggests that sorafenib may improve the efficacy of RFA.

DETAILED DESCRIPTION:
Hepatocellular cancer (HCC) has a poor prognosis with increasing mortality in the United States. Because HCC generally develops in patients with underlying liver disease, resection is often not possible. Liver transplant improves survival for HCC patients but given the national organ donor shortage often patients have to wait a considerable time for transplant. Liver-directed therapies such as radiofrequency ablation (RFA) remain important tools to control tumor growth and to potentially "bridge" patients to liver transplant. However, liver-directed therapies for HCC tumors greater than 3cm in size are suboptimal, leaving a critical unmet need.

Antiangiogenic systemic agents, such as oral sorafenib, reduce tumor blood flow and have been shown to improve RFA efficacy in animal and in computer models.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hepatocellular cancer (HCC) by pathology or by NCCN imaging guidelines
* All HCC stages are allowed. May be a liver transplant candidate.
* At least one tumor (index tumor) accurately measured as 3.5-7cm in diameter (long and short axis diameter to be recorded, but only one needs to meet this criteria) on baseline imaging.
* No prior therapy for the index tumor
* No prior systemic treatment for HCC within 4 weeks and no prior anti-VEGF therapy within 8 weeks of study entry.
* Life expectancy > 8 weeks.
* ECOG >=0 or 1
* RFA clinically indicated for index tumor.
* Acceptable overall RFA and anesthesia risk.
* Adequate bone marrow, liver and renal function: Hemoglobin >9.0 g/dl; Absolute neutrophil count (ANC)>1,500/mm3; Platelet count correctable to >50,000/mm3; compensated liver function (Child-Turcotte-Pugh A, B7 or B8); Creatinine <1.5 times ULN; INR correctable to <1.5.
* Ability to take oral medication and no evidence of impaired absorption.

Exclusion Criteria

* Urgent treatment of the index tumor anticipated.
* Participants who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Participants currently receiving any other study agents.
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib.
* Participants receiving medications or substances that are inducers of CYP3A4 (rifampicin, St. John's wort, phenytoin, carbamazepine, phenobarbital and dexamethasone) or that are metabolized/eliminated by predominantly UGT1A1 pathway or by CYP2B6 and CYP2C8.
* Decompensated liver disease
* Uncontrolled hypertension
* Thrombolic or embolic events within the past 6 months.
* Hemorrhage/bleeding event within 4 weeks
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence of severe or uncorrectable bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of study entry.
* Contraindication to or inability to undergo the RFA procedure,
* Contraindication to or inability to undergo imaging with MRI
* Uncontrolled intercurrent illness
* Individuals with a history of a different malignancy unless disease-free for at least 5 years and are deemed by the Investigator to be at low risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy

For additional inclusion/exclusion criteria details contact Study Site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bullock, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hakime A, Hines-Peralta A, Peddi H, Atkins MB, Sukhatme VP, Signoretti S, Regan M, Goldberg SN. Combination of radiofrequency ablation with antiangiogenic therapy for tumor ablation efficacy: study in mice. Radiology. 2007 Aug;244(2):464-70. doi: 10.1148/radiol.2442061005. PMID 17641366
- [Derived] Bockorny B, Bullock AJ, Abrams TA, Faintuch S, Alsop DC, Goldberg SN, Ahmed M, Miksad RA. Priming of Sorafenib Prior to Radiofrequency Ablation Does Not Increase Treatment Effect in Hepatocellular Carcinoma. Dig Dis Sci. 2022 Jul;67(7):3455-3463. doi: 10.1007/s10620-021-07156-2. Epub 2021 Jul 23. PMID 34297268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from June 2009 through August 2013.
Period: Overall Study
Arm/Group | Sorafenib | Placebo
Started | 10 | 10
Started Treatment | 9 | 10
Evaluable RFA | 7 | 8
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Intercurrent illness | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 66 (11) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Present Liver Cirrhosis [Count of Participants; unit: Participants] | 10 | 10 | 20
Present Portal Vein Thrombosis [Count of Participants; unit: Participants] | 1 | 5 | 6
Tumor Size - Short Axis [Mean (Standard Deviation); unit: centimeters] | 4.4 (1.3) | 4.4 (1.4) | 4.4 (1.3)
Tumor Size - Long Axis [Mean (Standard Deviation); unit: centimeters] | 4.9 (1.7) | 5.3 (1.3) | 5.1 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Coagulation Zone Diameter-Short Axis
Description: The size of the coagulation zone was determined on CT imaging obtained after RFA for the single index tumor.
Time Frame: Up to day 50 from study enrollment (target 30 days after RFA)
Population: The analysis population is comprised of all participants who completed treatment ending with day 10 RFA.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 9 | 9
millimeters | 36.0 (7.8) | 35.1 (8.8)

2. Primary Outcome: Coagulation Zone Diameter-Long Axis
Description: The size of the coagulation zone was determined on CT imaging obtained after RFA for the single index tumor.
Time Frame: Up to day 50 from study enrollment (target 30 days after RFA)
Population: The analysis population is comprised of all participants who completed treatment ending with RFA.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 9 | 9
millimeters | 42.4 (9.2) | 44.1 (7.8)

3. Primary Outcome: Coagulation Zone Volume
Description: The size of the coagulation zone was determined on CT imaging obtained after RFA for the single index tumor.
Time Frame: Up to day 50 from study enrollment (target 30 days after RFA)
Population: The analysis population is comprised of all participants who completed treatment ending with RFA.
Measure: Mean (Standard Deviation); unit: centimeters^3
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 9 | 9
centimeters^3 | 30.7 (24.6) | 30.5 (21.5)
Statistical Analysis 1: Comparison: Sorafenib vs Placebo; Assuming the two trial arms were independent, the standard deviation was 0.5cm for both arms and a sample size of 16 evaluable patients (8 per arm), the study had an 84% power at a 5% (two-sided) significance level to detect 0.8cm difference in ablation zone size. In order to allow a 20% drop-out rate, a total of 20 subjects were accrued; Test type: Superiority; p = .794, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Feasibility Rate
Description: Feasibility rate is defined as the percentage of participants completing radiofrequency ablation following 9 days of sorafenib or placebo therapy.
Time Frame: Up to day 14 since enrollment
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (90% Confidence Interval); unit: percentage of particpants
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 10 | 10
percentage of particpants | 90 [60.6 to 99.5] | 90 [60.6 to 99.5]

5. Secondary Outcome: Number of Treatment-Related Grade 1-4 Adverse Events (AEs) by Day 9
Description: AEs were assessed based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v3.0). The number of Grade 1-4 AEs with treatment attribution possibly, probably or definitely related up to day 9 of study drug treatment were counted for this outcome. Worst grade by patient within AE type was calculated. Participants could have multiple different AE types within a grade.
Time Frame: Day 9
Population: The analysis population is comprised of all treated participants.
Measure: Number; unit: adverse events
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 9 | 10
adverse events | 8 | 4

6. Secondary Outcome: Number of Treatment-Related Grade 1-4 Adverse Events (AEs) on Day of Radiofrequency Ablation (RFA)
Description: AEs were assessed based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v3.0). The number of Grade 1-4 AEs with treatment attribution possibly, probably or definitely related on day of RFA treatment were counted for this outcome. Worst grade by patient within AE type was calculated. Participants could have multiple AE types within a grade.
Time Frame: Up to day 14 (target day 10 RFA)
Population: The analysis population is comprised of all participants who completed treatment ending with RFA.
Measure: Number; unit: adverse events
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 9 | 9
adverse events | 5 | 4

7. Secondary Outcome: Number of Treatment-Related Grade 1-4 Adverse Events (AEs) One Month After Radiofrequency Ablation (RFA)
Description: AEs were assessed based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v3.0). The number of Grade 1-4 AEs with treatment attribution possibly, probably or definitely related one month after RFA treatment were counted for this outcome. Worst grade by patient within AE type was calculated. Participants could have multiple AE types within a grade.
Time Frame: Up to day 40 post RFA (target 30 days)
Population: The analysis population is comprised of all treated participants who were evaluable for AEs at day40.
Measure: Number; unit: adverse events
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 8 | 8
adverse events | 8 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected on treatment days 1-10 and the day 40 follow-up visit.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term. The analysis population is all treated patients (n=1 dropped out before starting treatment.
Groups:
- Sorafenib: Participants received a nine-day course of oral sorafenib 400 mg twice a day and radiofrequency ablation (RFA) on Day 10. Tumors in each group underwent RFA using a standard regimen (1 cm tip, 70 ± 2º C, 5 min).
  Sorafenib
  radiofrequency ablation
- Placebo: Participants received a nine-day course of placebo pills twice a day and radiofrequency ablation (RFA) on Day 10. Tumors in each group underwent RFA using a standard regimen (1 cm tip, 70 ± 2º C, 5 min).
  radiofrequency ablation
Arm/Group | Sorafenib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=9) | Placebo (N=10)
Leukocytes (Investigations) | 1 | 0
Lymphopenia (Investigations) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Bilirubin (Investigations) | 1 | 0
Liver, hemorrhage (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=9) | Placebo (N=10)
Abdomen, pain (Gastrointestinal disorders) | 3 | 3
Agitation (Psychiatric disorders) | 0 | 1
Alkaline phosphatase (Investigations) | 3 | 5
Allergic reaction (Immune system disorders) | 1 | 0
ALT, SGPT (Investigations) | 7 | 5
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 2
Ascites (non-malignant) (Gastrointestinal disorders) | 2 | 3
AST, SGOT (Investigations) | 8 | 8
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bicarbonate (Metabolism and nutrition disorders) | 1 | 0
Bilirubin (Investigations) | 5 | 4
Cardiac-other (Cardiac disorders) | 1 | 0
Chest/thoracic pain NOS (General disorders) | 1 | 1
Coagulation-other (Investigations) | 3 | 3
Cognitive disturbance (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Creatinine (Investigations) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 3
Distention/bloating, abdominal (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Edema limb (General disorders) | 2 | 3
Edema trunk/genital (General disorders) | 0 | 1
Endocrine-other (Endocrine disorders) | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 3
Fever w/o neutropenia (General disorders) | 0 | 2
GI-other (Gastrointestinal disorders) | 2 | 3
Head/headache (Nervous system disorders) | 0 | 2
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 0 | 1
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 0 | 2
Hearing-other (Ear and labyrinth disorders) | 0 | 1
Hematologic-other (Blood and lymphatic system disorders) | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 4 | 3
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypertension (Vascular disorders) | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Incontinence urinary (Renal and urinary disorders) | 1 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1 | 0
INR (Investigations) | 5 | 5
Insomnia (Psychiatric disorders) | 1 | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Leukocytes (Investigations) | 3 | 1
Liver, hemorrhage (Hepatobiliary disorders) | 2 | 0
Liver, pain (Hepatobiliary disorders) | 1 | 0
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 2 | 0
Lymphopenia (Investigations) | 1 | 0
Metabolic/Laboratory-other (Investigations) | 2 | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Neuropathy-motor (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 2
Neutrophils (Investigations) | 3 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Ocular-other (Eye disorders) | 0 | 1
Oral cavity, pain (Gastrointestinal disorders) | 1 | 0
Pain-other (General disorders) | 2 | 3
Palpitations (Cardiac disorders) | 0 | 1
Pancreatic glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Peritoneal cavity, hemorrhage (Gastrointestinal disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Platelets (Investigations) | 7 | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 | 1
PTT (Investigations) | 1 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Renal/GU-other (Renal and urinary disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 2
Stomach, pain (Gastrointestinal disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 1
Teeth (Gastrointestinal disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Urethra, pain (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Varices (rectal), hemorrhage (Gastrointestinal disorders) | 1 | 1
Viral hepatitis (Infections and infestations) | 1 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 3 | 2

LIMITATIONS AND CAVEATS:
This study is limited by small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No